CLINICAL TRIAL: NCT03576482
Title: Emotional Impact of the Way Conducting Cancer Patients to the Surgical Center: a Randomized Clinical Trial Comparing Transport by Stretcher on Wheels and Ambulation.
Brief Title: Emotional Impact of the Way Conducting Cancer Patients to the Surgical Center
Status: Completed | Type: Observational
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ricardo dos Reis, PhD, Barretos Cancer Hospital
Other Study IDs: 1527/2018
Record Dates: First submitted 2018-06-13; First posted 2018-07-03 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Anxiety Disorders; Depression
Keywords: Anxiety disorders; Depression; Transport to operating room
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transport on foot: Patients go to operating room walking with their families and with their normal clothes
  Interventions: Other: Transport on foot
- Transport by stretcher on wheels: Patients go to operating room by stretcher on wheels and with hospital clothes. Normal routine of our hospital.

INTERVENTIONS:
Other: Transport on foot — Patients go to operating room walking with their families and with their normal clothes
  Groups: Transport on foot

SUMMARY:
Cancer is an extremely aggressive disease, anxiety and depression are consequences some patients may develop from diagnosis continuing during treatment. A measures control of the cancer is surgery for removal tumor. The surgical procedure is often a difficult experience for patients and their relatives, and patients in the preoperative period are often psychological symptoms of anxiety and depression. A previous study with the objective analyzing patient's emotional repercussion according the type of transport to the surgical center reached the following result: patients who go to the surgical center feel more relaxed in the preoperative period.

The primary objective is to analyze emotional repercussion of patient diagnosed with cancer classified in Eastern Cooperative Oncology Group (ECOG) Performance Status 0 and 1 according type transport to the surgical center.

DETAILED DESCRIPTION:
A randomized clinical trial, prospective collection to be performed at the Barretos Cancer Hospital, will be include 176 patients, 88 patients being allocated to transport to operating room by stretcher on wheels (group 1) and 88 patients being allocated to transport to operating room by ambulation (group 2). Patients with indication elective surgery that meet the inclusion criteria will be included, and randomized for one of the groups, and may be referred by stretcher on wheels to the surgical center (group 1) or referred to the surgical center by ambulation (group 2). The Hospital Anxiety and Depression Scale (HAD) and the survey developed for the present study Sati-Cir, Evaluation Questionnaire of Satisfaction with Healthcare in Surgery, will be the instruments used in data collection. Participants will respond both after the course to the surgical center.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed cancer
* Age ≥18 years, ≤ 70 years
* Both sexes
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score 0 or 1
* Patients classified as Zero or Low Risk by the fall risk assessment scale
* Indication elective surgery

Exclusion Criteria:

* Patients who present moments before surgery has an adverse event that could jeopardize the ambulation to the surgical center.
* Patients who are physically disabled and require assistance walking.
* Patients has indication bed in the Intensive Care Unit (UTI)
* Patients has previously diagnosed psychiatric disorders (severe depression, anxiety disorder, panic, among others).
* Patients doens't have an accompanying person on the day of surgery.
* Patients taking anxiolytic and antidepressant medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be organized including 176 patients sheduled for elective cancer surgery at Barretos Cancer Hospital, 88 patients bei ng allocated for transporting to the operating room by stretcher on wheels, and 88 patients elective allocated for transporting to the operating room by ambulation.
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression levels | up to 4 weeks
  Measure the anxiety and depression levels using Hospital Anxiety and Depression Scale (HAD) and the survey developed for the present study Sati-Cir, Evaluation Questionnaire of Satisfaction with Healthcare in Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela da S Oliveira, Nurse, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Hospital do Câncer de Barretos, Barretos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We do not intend to share our individual participant data to other researches

REFERENCES:
- [Derived] Oliveira GDS, Sabaini PMDS, Pedrao PG, da Silva VB, Lima MA, Mantovani TEDS, Andrade CEMDC, Dos Reis R. Emotional impact according to the way cancer patients are conducted to the surgical center: A randomized clinical trial comparing ambulation to the stretcher. PLoS One. 2025 Apr 22;20(4):e0320856. doi: 10.1371/journal.pone.0320856. eCollection 2025. PMID 40261947